CLINICAL TRIAL: NCT05491330
Title: Comparative Randomized, Single Dose, Three-way, Three-sequence, Two Treatment, Partial Replicate, Crossover, Open-label Study to Determine the Bioequivalence of Nirmatrelvir & Ritonavir From Copaxid 150 +100 mg Tablets (Eva Pharma, Egypt) Versus Paxlovid 150 + 100 mg Film Coated Tablets (Pfizer Europe, Belgium)
Brief Title: Bioequivalence Study of Nirmatrelvir & Ritonavir From Copaxid 150 +100 mg Tablets (Eva Pharma, Egypt) Versus Paxlovid 150 + 100 mg Film Coated Tablets (Pfizer Europe, Belgium)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genuine Research Center, Egypt (Industry)
Collaborators: Eva Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: GRC/1/22/1038
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Healthy
MeSH Terms: interventions — nirmatrelvir; Ritonavir; nirmatrelvir and ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- R reference (first dose) (Active Comparator): Reference drug (Paxlovid) Nirmatrelvir 150 mg + Ritonavir 100 mg tablets
  Interventions: Drug: Nirmatrelvir 150 mg + Ritonavir 100 mg (Reference first dose)
- T test (Experimental): Test drug (Copaxid) Nirmatrelvir 150 mg + Ritonavir 100 mg tablets
  Interventions: Drug: Nirmatrelvir 150 mg + Ritonavir 100 mg (test)
- R reference (second dose) (Active Comparator): Reference drug (Paxlovid) Nirmatrelvir 150 mg + Ritonavir 100 mg tablets
  Interventions: Drug: Nirmatrelvir 150 mg + Ritonavir 100 mg (Reference second dose)

INTERVENTIONS:
Drug: Nirmatrelvir 150 mg + Ritonavir 100 mg (Reference first dose) — 2 tablets from Nirmatrelvir 150 mg + 1 tablet from Ritonavir 100 mg
  Other Names: Paxlovid
  Arms: R reference (first dose)
Drug: Nirmatrelvir 150 mg + Ritonavir 100 mg (test) — 2 tablets from Nirmatrelvir 150 mg + 1 tablet from Ritonavir 100 mg
  Other Names: Copaxid
  Arms: T test
Drug: Nirmatrelvir 150 mg + Ritonavir 100 mg (Reference second dose) — 2 tablets from Nirmatrelvir 150 mg + 1 tablet from Ritonavir 100 mg
  Other Names: Paxlovid
  Arms: R reference (second dose)

SUMMARY:
Comparative randomized, single dose, three-way, three-sequence, two treatment, partial replicate, crossover, open-label study to determine the bioequivalence of Nirmatrelvir & Ritonavir From Copaxid 150 +100 mg Tablets (Eva Pharma, Egypt) Versus Paxlovid 150 + 100 mg Film Coated Tablets (Pfizer Europe, Belgium)

DETAILED DESCRIPTION:
Primary Pharmacokinetic Parameters: Cmax, AUC0→t and AUC0→∞ Secondary Pharmacokinetic Parameters: Ke, tmax and t1/2e. ANOVA using 5% significance level for transformed (with the 90% confidence intervals) and untransformed data of Cmax, AUC0→t and AUC0→∞ and for untransformed data of Ke, tmax and t1/2e.

The confidence intervals of logarithmically transformed Test/Reference ratios for Cmax, AUC0→t and AUC0→∞ to be within 80.00-125.00%.

A comprehensive final report will be issued upon the completion of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female, age 18 to 55 years, inclusive.
2. Body weight within 15% of normal range according to the accepted normal values for body mass index (BMI).
3. Medical demographics without evidence of clinically significant deviation from normal medical condition, eg.: no history of heart, liver, kidney, gastrointestinal, nervous system, or metabolic abnormalities.
4. Results of clinical laboratory test are within the normal range or with a deviation that is not considered clinically significant by principal investigator.
5. Females should be on a suitable birth control method.
6. Fully informed subjects that consented to participate in the study.

Exclusion Criteria:

1. Subjects with known allergy to the products tested.
2. Female subjects who were pregnant or nursing.
3. Acute infection within one week preceding first study drug administration.
4. History of drug or alcohol abuse.
5. Subject does not comply with the stated instruction of not taking any prescription or non-prescription drugs within two weeks before first study drug administration and until the end of the study.
6. Subject is on a special diet (for example subject is vegetarian).
7. Subject does not agree not to consume any beverages or foods containing methyl-xanthenes e.g. caffeine (coffee, tea, cola, chocolate etc.) 48 hours prior to the study administration of either study period until donating the last sample in each respective period.
8. Subject does not agree not to consume any beverages or foods containing grapefruit 7 days prior to first study drug administration until the end of the study.
9. Subject has a family history of severe diseases which have direct impact on the study.
10. Participation in a bioequivalence study or in a clinical study within the last 8 weeks before first study drug administration.
11. Subject intends to be hospitalized within 3 months after first study drug administration.
12. Subjects who have donated blood or lost more than 500 mL blood within 3 months prior to the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2022-08-21 (Actual); Primary Completion 2022-09-04 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
Cmax | Up to 48 hours post dose in each treatment period
  Maximal measured plasma concentration

SECONDARY OUTCOMES:
Time of the maximum plasma concentration (Tmax) | Up to 48 hours post dose in each treatment period
  The amount of time that a drug is present at the maximum concentration in serum

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elshafeey, Ph.D. Pharma, Study Director — Genuine Research Center
Locations (1):
- Genuine Research Center GRC, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chow SC, Wang H. On sample size calculation in bioequivalence trials. J Pharmacokinet Pharmacodyn. 2001 Apr;28(2):155-69. doi: 10.1023/a:1011503032353. PMID 11381568
- [Background] Diletti E, Hauschke D, Steinijans VW. Sample size determination for bioequivalence assessment by means of confidence intervals. Int J Clin Pharmacol Ther Toxicol. 1991 Jan;29(1):1-8. PMID 2004861
- [Background] Schuirmann DJ. A comparison of the two one-sided tests procedure and the power approach for assessing the equivalence of average bioavailability. J Pharmacokinet Biopharm. 1987 Dec;15(6):657-80. doi: 10.1007/BF01068419. PMID 3450848